CLINICAL TRIAL: NCT00505362
Title: Rectus Muscle Closure vs. Non-Closure at Primary Cesarean Delivery and Post-Operative Pain
Brief Title: Pain Study of Rectus Muscle Closure at Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Deirdre Judith Lyell, Associate Professor of Obstetrics and Gynecology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6107
Record Dates: First submitted 2007-07-19; First posted 2007-07-23 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rectus muscle closure (Active Comparator): Two-layer uterine closure, peritoneal closure, fascial and skin closure and reapproximation of the rectus muscles with three-interrupted sutures.
  Interventions: Procedure: Rectus closure
- Rectus muscle non-closure (No Intervention): Two-layer uterine closure, peritoneal closure, fascial and skin closure, and rectus muscles non-closure.

INTERVENTIONS:
Procedure: Rectus closure — Reapproximation of the rectus muscles with three-interrupted sutures
  Arms: Rectus muscle closure

SUMMARY:
Suture reapproximation of the rectus muscles at primary cesarean delivery is a common practice about which there are no data. Some Obstetricians believe that suture reapproximation of the rectus muscles increases post-operative pain, and it may decrease adhesions, yet there are no published data to support or refute these claims. The purpose of this study is to assess the effect of rectus muscle reapproximation at cesarean delivery and post-operative pain. We also plan to assess the impact of rectus muscle closure on adhesions as seen at repeat cesarean delivery.

DETAILED DESCRIPTION:
There are more than 1 million cesarean deliveries performed annually in the United States, at a rate of 30.2% of all deliveries. Data are limited regarding optimal surgical closure techniques to minimize adhesions at cesarean. Adhesions are implicated in pelvic pain, infertility, difficult repeat surgery, and bowel obstruction. Practice techniques regarding rectus muscle reapproximation vary widely, and there are no data regarding the impact of this step on pain, and some data suggesting a reduction in significant adhesions. Given the frequency of cesarean deliveries, small changes in surgical technique may yield significant benefits.

We hope to learn 1) whether suture reapproximation of the rectus muscles increases pain, and 2) the degree to which suture reapproximation of the rectus muscles alters adhesions when studied in a prospective, randomized trial.

All patients undergoing primary cesarean delivery at Lucile Packard Childrens Hospital (LPCH) will be offered the study. Once consented, patients will be randomized to one of two standardized closure techniques at cesarean: two-layer uterine closure, peritoneal closure, fascial and skin closure, and either reapproximation of the rectus muscles with three-interrupted sutures, or non-closure. Intra-operative and post-operative pain management will be standardized. Subjects will undergo pain assessments while in-house on post-operative days 1 and 3, and at the standard post-partum clinic visit after 6 weeks. These assessments will require less than 5 minutes of the patient's time. Patients will be shown a pain chart, and will be asked to rate their pain on a scale of 0 to 10 at rest. They will then stand up and rate their pain again. Pain medication usage will also be assessed.

The surgeons will know the groups to which the patients are randomized. The patients and those collecting data on pain scores will not.

Primary Endpoint: combined opioid use and movement pain score (Silverman Integrated Assessment-SIA) 72 post-operative hours.

Secondary Endpoint: surgical complications, maternal satisfaction with analgesia.

ELIGIBILITY:
Inclusion Criteria:

37 weeks gestation Primary cesarean American Society of Anesthesiologists (ASA) class 1 or class 2

Exclusion Criteria:

Chronic analgesia use Vertical skin incision at cesarean Opioid or Non-steroidal anti-inflammatory drugs (NSAID) allergy BMI >40 Labor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2006-06; Primary Completion 2014-08 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Judith Lyell, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rectus Muscle Closure | Rectus Muscle Non-closure
Started | 35 | 28
Completed | 35 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rectus Muscle Closure | Rectus Muscle Non-closure | Total
Number analyzed (Participants) | 35 | 28 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (7) | 33 (7) | 32 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 28 | 63
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 28 | 63
Gestational age at delivery [Median (Inter-Quartile Range); unit: weeks] | 39 [37 to 39] | 38 [37 to 39] | 39 [37 to 39]

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain
Description: Post-operative pain was assessed using Silverman Integrated Assessment (SIA) pain score which combines the opioid use and movement pain score over the 72-hour study period. The SIA pain and opioid score is calculated by first rank ordering each patient's total opioid use (morphine milligram equivalents) and area under the curve (AUC) movement pain score over the 72 hour study period, then calculating a mean for both opioid use and movement pain scores, expressing both opioid use and movement pain score as percent differences from the mean, and lastly adding the percent differences from the mean for the two variables. The SIA composite score value for each subject ranges from approximately 200% to approximately -200%, with the highest positive score indicating the least comfortable or the most pain despite the greatest use of analgesics, and the lowest score indicating the most comfortable or least pain despite the least use of analgesics.
Time Frame: 72-hour study period
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Rectus Muscle Closure | Rectus Muscle Non-closure
Number analyzed (Participants) | 35 | 28
Scores on a scale | 15 (100) | -31 (78)
Statistical Analysis 1: Comparison: Rectus Muscle Closure vs Rectus Muscle Non-closure; Test type: Superiority or Other; p = 0.04, t-test, 2 sided

2. Secondary Outcome: Operative Times
Description: Operative time of the cesarean delivery in minutes.
Time Frame: From start to the end of the cesarean delivery, assessed up to two hours.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Rectus Muscle Closure | Rectus Muscle Non-closure
Number analyzed (Participants) | 35 | 28
minutes | 63 (15) | 65 (15)
Statistical Analysis 1: Comparison: Rectus Muscle Closure vs Rectus Muscle Non-closure; Test type: Superiority or Other; p = 0.61, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 weeks after the delivery
Arm/Group | Rectus Muscle Closure | Rectus Muscle Non-closure
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/28
Other Adverse Events (participants affected / at risk) | 0/35 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No